CLINICAL TRIAL: NCT03993548
Title: KickStart30: A 30-Day Intervention for Patients With Rheumatoid Arthritis (RA)
Acronym: KickStart30
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Saundra Jain, Adjunct Clinical Affiliate, School of Nursing, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-10-0095
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-03

CONDITIONS: Chronic Pain; Stress; Psychological; Healthy; Rheumatoid Arthritis
Keywords: Wellness; Mental Wellness; Well-Being
MeSH Terms: conditions — Chronic Pain; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wellness Intervention (Experimental): KickStart30 is an integrated, prescriptive, and trackable wellness intervention combining five wellness elements including exercise, mindfulness, sleep, social connectedness, and nutrition.
  Interventions: Behavioral: Wellness Element 1 - Exercise; Behavioral: Wellness Element 2 - Mindfulness; Behavioral: Wellness Element 3 - Sleep Hygiene; Behavioral: Wellness Element 4 - Social Connectedness; Behavioral: Wellness Element 5 - Nutrition; Behavioral: Wellness Element 6 - Wellness Exercises; Behavioral: Wellness Element 7 - Motivational Messages

INTERVENTIONS:
Behavioral: Wellness Element 1 - Exercise — Daily wellness element focusing on Exercise; adherence documented online daily
Behavioral: Wellness Element 2 - Mindfulness — Daily wellness element focusing on Mindfulness Meditation; adherence documented online daily
Behavioral: Wellness Element 3 - Sleep Hygiene — Daily wellness element focusing on sleep hygiene; adherence documented online daily
Behavioral: Wellness Element 4 - Social Connectedness — Daily wellness element focusing on Social Connectedness; adherence documented online daily
Behavioral: Wellness Element 5 - Nutrition — Daily wellness element focusing on Nutrition; adherence documented online daily
Behavioral: Wellness Element 6 - Wellness Exercises — Daily wellness workbook exercises focusing on improving mental wellness; adherence documented online daily
Behavioral: Wellness Element 7 - Motivational Messages — Daily motivational emails offering information on one of the 5 wellness elements each day (Exercise, Mindfulness Meditation, Sleep, Social Connectedness, and Nutrition)

SUMMARY:
This study explores the efficacy and feasibility of a self-management wellness intervention that is integrated, prescriptive, and trackable in a population of patients with Rheumatoid Arthritis (RA) taking a biologic. This 30-day wellness intervention (called "KickStart30") combines five wellness elements: exercise, mindfulness, sleep, social connectedness, and nutrition. Additionally, the program requires that participants implement 5 wellness interventions daily for the 30-day study, document daily online adherence, complete daily HERO (happiness, enthusiasm, resilience, and optimism) exercises to improve mental wellness, and complete online program forms before and after the 30-day intervention. Participants are assessed pre- and post-intervention to determine whether the intervention promotes wellness behavior changes.

DETAILED DESCRIPTION:
It is expected that this 30-day integrated, prescriptive, and trackable wellness intervention (combining five wellness elements including exercise, mindfulness, sleep, social connectedness, and nutrition) will be found to be an efficacious program for those with Rheumatoid Arthritis taking a biologic or a JAK inhibitor.

Traditionally mental health and other specialties like rheumatology have focused primarily on the diagnosis and treatment of illness rather than incorporating wellness as an essential element of treatment. Those in the helping professions are trained to diagnose health problems with treatment typically focusing on symptom reduction. More recently, mental health and other healthcare specialties like rheumatology have initiated a conversation and subsequent research focusing on the importance of integrating elements of wellness into treatment. Rather than focusing solely on symptom reduction, some providers have begun incorporating elements of wellness promotion into treatment with favorable results.

To the best of our knowledge, even though there is abundant research supporting each of the KickStart30 elements (exercise, mindfulness, sleep, social connectedness, and nutrition) individually, there is no research exploring the effectiveness of an integrated, prescriptive, and trackable wellness intervention combining these five elements specific to a cohort of patients with RA. Therefore, this work will be unique in that it will collect both objective and subjective data to assess the feasibility and effectiveness of this type of wellness intervention. It will lend support to the growing body of research on the efficacy of wellness interventions for a variety of different health conditions, as well as a community-based population. Finally, it is hoped that positive results will yield increased access to and utilization of this type of intervention, thereby improving public health.

The recruitment period will be open for 12 months to obtain a maximum of 50 participants. The study population will be individuals, ages 18 and older, interested in improving their overall wellness and that self-identify as having Rheumatoid Arthritis and taking a biologic or a JAK inhibitor. Each participant will be engaged in the program for 30 days. To determine a participant's eligibility, study personnel will conduct a preliminary screening/orientation telephone interview. If the participant is determined to be eligible for the study based on the preliminary screening/orientation phone interview, study personnel will collect the participant's email address, physical mailing address, and assign the participant a unique identification code based on the order in which the participant was screened. The consent form outlines the purpose and design of the study, data to be collected, confidentiality standards, alternatives to participation, and contact information for research personnel. Participants will have the option to download a PDF of their signed consent form for their records at the time of signing/completion.

Study personnel will mail each participant a KickStart30 Workbook within one day of emailing participants their unique identification codes. Participants will be instructed to document adherence of their daily wellness practices and their daily HERO exercises online via Qualtrics, an online survey software. Participants can document their daily adherence using their computer and/or their smartphone as Qualtrics offers a mobile version of the Participant Tracking Form. A copy of the Participant Tracking Form will also be available in the KickStart30 Workbook so participants that prefer keeping a daily paper log can do so, and they can then transfer their program adherence information to the online Participant Tracking Form at their convenience throughout the program. The workbook will contain the participant's personal identification code; no personal identification will appear in the workbook in order to protect participant confidentiality. Participants will also receive daily motivational emails from MailChimp, which will provide general information about one of the five wellness elements and/or one of the HERO wellness traits, as well as encouragement to track their participation on a daily basis, and encouragement to contact study personnel via email with any questions and/or concerns.

Data capture will occur at two points: once prior to beginning the study and again at the end of the 30-day study. Data will be collected online through program forms; all data will be hosted on Qualtrics, an online survey software. Program Forms assess items including depression, anxiety, wellbeing, mindfulness, sleep quality, social connectedness, emotional eating, pain, disability, physical function, happiness, enthusiasm, resilience, and optimism in patients with RA.

Descriptive statistics will be used to discuss pre- and post-intervention scores. Differences between pretest and 30-day measures will be assessed with repeated measures ANOVA, with a p value of less than 0.05 indicating statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Rheumatoid Arthritis (RA) by a Rheumatologist
* Currently taking a biologic and/or a JaK inhibitor for the treatment of RA, including one or more of the following: Orencia (intravenous infusion or subcutaneous injection), Humira (subcutaneous injection), Kineret (subcutaneous injection), Cimzia (subcutaneous injection), Enbrel (subcutaneous injection), Simponi (subcutaneous injection), Simponi Aria (intravenous infusion), Remicade (intravenous infusion), Kevzara (subcutaneous injection), Rituxan (intravenous infusion), Actemra (intravenous infusion or subcutaneous injection), Olumiant (oral administration), Xeljanz (oral administration)
* Interested in improving overall wellness
* Not pregnant and no plans to get pregnant during the 30-day study
* English-speaking
* Must have access to a reliable Internet-enabled computer
* Must possess basic computer skills

Exclusion Criteria:

* Has not been diagnosed with RA by a Rheumatologist
* Not currently taking a biologic or a JAK inhibitor for the treatment of RA
* Not interested in improving overall wellness
* Pregnant or plans to get pregnant during the 30-day study
* Does not speak English
* Does not have access to a reliable, Internet-enabled computer
* Reports a lack of basic computer skills
* Acutely suicidal and/or actively psychotic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) | 0, and 30 days
  The PHQ-9 is a nine-item depression self-report questionnaire for screening and measurement of severity of major depression. Scores range from 0-27 (Lower scores = Less depression).
Change in Generalized Anxiety Disorder-7 (GAD-7) | 0, and 30 days
  The GAD-7 is a seven-item self-report questionnaire for screening and measurement of severity of generalized anxiety disorder. Scores range from 0-21 (Lower scores = Less anxiety).
Change in World Health Organization Well-Being Index (WHO-5) | 0, and 30 days
  The WHO-5 Well-Being Index is a five-item self-report questionnaire covering 5 areas: positive mood, vitality, and general interests. Scores range from 0-25 (Higher scores = Higher levels of well-being).
Change in Mindful Attention Awareness Scale (MAAS) | 0, and 30 days
  The MAAS is a 15-item scale designed to assess a core characteristic of dispositional mindfulness. Scores range from 15-90 (Higher scores = Higher levels of mindfulness).
Change in Sleep Condition Indicator (SCI) | 0, and 30 days
  The SCI is a brief 8-item screening tool to evaluate insomnia disorder. Scores range from 0-32 (Lower scores = Greater sleep problems).
Change in Social Connectedness Scale (SCS) | 0, and 30 days
  The SCS is an 8-item questionnaire that assesses the degree to which people feel connected to others in their social environment. Scores range from 8 to 48. (Higher scores = More connectedness to others).
Change in Eating and Appraisal Due to Emotions and Stress (EADES) | 0, and 30 days
  The EADES is a 24-item sub-scale used to measure stress-related eating. Scores range from 24-120 (Lower scores = Greater emotion and stress-related eating).
Change in Brief Pain Inventory (BPI) | 0, and 30 days
  The BPI is an 8-item scale that assesses pain. Scores range from 0-10. (0 = No pain and 10 = Pain as bad as you can imagine).
Change in Sheehan Disability Scale (SDS) | 0, and 30 days
  The SDS is a 3-item measurement tool for assessing functional impairment in three inter-related domains: work/school, social, and family life. Scores range from 0-10 (Higher scores = Higher levels of functional impairment).
Change in Cognitive and Physical Functioning Questionnaire (CPFQ) | 0, and 30 days
  The CPFQ is a brief 7-item scale designed to assess cognitive and physical functioning. Scores range from 7-42 (Lower scores = Higher levels of cognitive and physical functioning).
Change in HERO Wellness Scale | 0, and 30 days
  The HERO Wellness Scale is a brief 5-item scale designed to measure four wellness traits plus perceived mental wellness. Scores range from 0-50 (Lower scores = Lower levels of mental wellness).
Post-Program Participant Questionnaire | 0, and 30 days
  A brief 6 question post study survey that captures participants' opinions about KickStart30.
Change in Health Assessment Questionnaire-II (HAQ-II) | 0, and 30 days
  The HAQ-II is a ten-item self-report questionnaire for assessing functional status in individuals with rheumatic disease. Scores range from 0-3.0 (Higher scores = Worse functioning and greater disability).

CONTACTS AND LOCATIONS:
Overall Officials: Saundra M Jain, PsyD, LPC, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No